CLINICAL TRIAL: NCT04192578
Title: The Effect of Remote Ischemic Conditioning on 2,3-bisphosphoglycerate in Erythrocyte
Brief Title: Effect of RIC on 2,3-BPG in Erythrocyte (RIC-BPG)
Acronym: RIC-BPG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RIC-2,3-BPG
Record Dates: First submitted 2019-10-31; First posted 2019-12-10 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: 2,3-Bisphosphoglycerate
Keywords: Remote ischemic conditioning; 2,3-Bisphosphoglycerate; Erythrocyte; Oxygen; healthy subjects

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Unilateral upper limb 60mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on unilateral upper limb and inflated to 60 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning
- Bilateral upper limb 60mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on bilateral upper limb and inflated to 60 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning
- Unilateral upper limb 200mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on unilateral upper limb and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning
- Bilateral upper limb 200mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on bilateral upper limb and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning
- Unilateral lower limb 60mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on unilateral lower limb and inflated to 60 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning
- Bilateral lower limb 60mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on bilateral lower limb and inflated to 60 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning
- Unilateral lower limb 200mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on unilateral lower limb and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning
- Bilateral lower limb 200mmHg RIC (Experimental): RIC is a physical strategy performed by an electric autocontrol device with cuffs placed on bilateral lower limb and inflated to 200 mmHg for 5-min followed by deflation for 5-min, the procedures is performed repeatedly for 5 times.
  Interventions: Device: remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — RIC is induced by short-term insulting blood-flow of nonvital distant organs intermittently.

SUMMARY:
Under hypoxia or high-altitude hypoxia ,it has been found that 2,3-bisphosphoglycerate(2,3-BPG) in erythrocyte increased and facilitated oxygen release to tissues.Remote Ischemic Conditioning(RIC) can also cause hypoxic conditions in local limbs.Thus,we hypothesize that whether RIC could also increase 2,3-BPG in erythrocyte.

DETAILED DESCRIPTION:
RIC is induced by short-term insulting blood-flow of nonvital distant organs intermittently and has been proved to be effective in ischemic stroke and myocardial infarction(MI).The possible mechanisms of RIC protection is complicated.RIC leads to local ischemia and hypoxia and has been demonstrated to play a role in vital organs through hypoxia inducible factors(HIF) against stroke and MI.Besides HIF, hypoxia or high-altitude hypoxia could also change glycolytic process in erythrocyte through adenosine or sphingosine-1-phosphate(S1P).Accompanying with alternating glucolysis, 2,3-diphosphoglycerate(2,3-BPG) in erythrocyte increases and it also facilitating oxygen release to tissues.Thus,we hypothesize that whether RIC could also increase 2,3-BPG in erythrocyte.There are 8 arms in this trial: All arms are RIC treatment. The level of 2,3-BPG in erythrocyte will be assessed by ELISA before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-65 years old
2. Healthy adults

Exclusion Criteria:

1. Individuals with various chronic diseases.
2. Individuals with various acute diseases.
3. Individuals who take any medicines
4. Individuals who have taken health supplements for more than 2 weeks.
5. individuals with BMI<18.5 or BMI≥24

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes of 2,3-BPG levels in erythrocyte | through study completion, an average of 24 hours
  Whole blood for testing effect of RIC on 2,3-BPG in Erythrocyte

SECONDARY OUTCOMES:
Changes of prothrombin time(PT) | through study completion, an average of 24 hours
  Whole blood for testing effect of RIC on PT
Changes of activated partial thromboplastin time(APPT) | through study completion, an average of 24 hours
  Whole blood for testing effect of RIC on APPT
Changes of activated partial thrombin time(TT) | through study completion, an average of 24 hours
  Whole blood for testing effect of RIC on TT
Changes of Fibrinogen(FIB) | through study completion, an average of 24 hours
  Whole blood for testing effect of RIC on FIB
Changes of D-dimer | through study completion, an average of 24 hours
  Whole blood for testing effect of RIC on D-dimer
Changes of hypoxia inducible factor-1(HIF-1) | through study completion, an average of 24 hours
  Whole blood for testing effect of RIC on HIF-1
Changes of lower limbs venous blood flow | through study completion, an average of 24 hours
  Vascular ultrasound for detecting venous blood flow in lower limbs

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, PhD, Principal Investigator — Xuanwu Hospital, Beijing